CLINICAL TRIAL: NCT06741371
Title: Impact of Using Synthetic Absorbable Monofilament Versus Multifilament Suture Material for Uterine Closure on the Development of Uterine Isthmocele : A Rondamized Controlled Clinical Trial
Brief Title: Difference Between Monofilament Versus Multifilament Suture Material in Isthmocele Formation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohammed Essam ElDin Mohammed, Assistant lecturer, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU MD333/2023
Record Dates: First submitted 2024-12-08; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Uterine Scar
MeSH Terms: interventions — glycolide E-caprolactone copolymer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monocryl arm (Experimental)
  Interventions: Procedure: Monocryl
- Vicryl arm (No Intervention)

INTERVENTIONS:
Procedure: Monocryl — Closure of the uterine scar by monofilament suture material
  Arms: Monocryl arm

SUMMARY:
This thesis conducts the effect of using different suture materials on the development of uterine scar niche after cesarean section.

The difference between monofilament and multifilament sutures and the special properties of each one .

The primary outcome of the study is to know which material conducts more scar niche formation .

Secondary outcomes are the extent of blood loss , the need of extra hemostatic sutures

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-45 years old

  * Singleton pregnancy.
  * Gestational age between 37 completed weeks to 42 weeks.
  * Patients undergoing elective primary caesarean section

Exclusion Criteria:

* History of uterine surgery (e.g. hysterotomy, myomectomy, perforation, caesarean section). (to be able to differentiate between the recent CS scar and the old scar)

  * Abnormal placental invasion (placenta previa and accrete ) ( more liable to undergo Cesarean hysterectomy)
  * Uterine anomalies (e.g., septum, Mullerian anomalies or fibroids). (may be localized at the suture line and therefore affect the scar)
  * Drugs intake that affects bleeding or tissue healing e.g., anti-coagulants, immunosuppressive drugs and chronic use of steroids (more than 14 days pre-operative)
  * Any medical Co-morbidity (diabetes mellitus, Hypertension and Thyroid abnormalities) (more liable to affect the healing)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of isthmocele by transvaginal ultrasound 6 months after delivery | 6 months
  Effect of using monofilament sutures on the development of uterine scar niche

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT06741371/Prot_ICF_000.pdf